CLINICAL TRIAL: NCT05810779
Title: Comparison of Dynamic Surface Exercise and Trunk Targeted Training on Gross Motor Function, Balance and Trunk Control in Children With Spastic Cerebral Palsy
Brief Title: Dynamic Surface Exercise and Trunk Targeted Training in Children With Spastic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0742
Record Dates: First submitted 2023-01-04; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Spastic Cerebral Palsy
Keywords: Balance; Cerebral palsy; Dynamic surface training; Gross motor function.
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dynamic surface exercise with conventional therapy (Experimental): the experimental group undergo conventional physical therapy and additional dynamic surface exercise training thrice a week for 2 months dynamic surface training will include gym balls , bolster or platform swing
  Interventions: Other: dynamic surface exercise
- trunk targeted training with conventional therapy (Active Comparator): the group will receive conventional physical therapy and additional trunk targeted training thrice a week for 2 months.
  Interventions: Other: trunk targeted training

INTERVENTIONS:
Other: dynamic surface exercise — Optimal arousal Physio ball Make the child bounce, active/passive on the Swiss ball, slow/fast 5 times 5 sets Combined frontal and transverse plane movements Physio ball/ bolster High sitting: one hand weight bearing followed by trunk rotation to reach the toy on opposite side 5-7 each side 1 set Combined frontal and transverse plane movements Platform swing Reaching the toy with both the hands kept overhead and 45°-60° diagonal to the mid line 5-7 times each side 1 set
  Other Names: comparison between dynamic surface exercise and trunk targeted training
  Arms: dynamic surface exercise with conventional therapy
Other: trunk targeted training — trunk training group (TTG) consist of exercises and activities focusing on the activation of the trunk muscles, pelvic control and proximal stabilization and these were combined with the trunk and gluteal muscle strengthening exercises.
  The trunk elongation activities, the facilitation of spinal extension, weight shifting and weight-bearing activities The children in the TTG received 45-75-minute of physiotherapy twice a week for 8 weeks
  Other Names: comparison between dynamic surface exercise and trunk targeted training
  Arms: trunk targeted training with conventional therapy

SUMMARY:
This study aims to describe the comparative effects of dynamic surface training and trunk targeted training in order to ensure which method is best in improving gross motor function , balance and trunk control in children with spastic cerebral palsy . this will be randomized control study which includes participants with age 5 to 10 years

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a well-documented nonprogressive neurodevelopmental condition commencing in early childhood and persisting throughout life. The neuromuscular deficits observed in children with CP include abnormal muscle tone that affects posture, movement, alteration of balance and motor coordination, decrease in strength, and loss of selective motor control, leading to functional limitation. Neurodevelopmental principles state that the control of movement proceeds from the proximal to the distal part of the body. The trunk being the central key point of the body, proximal trunk control is a prerequisite for distal limb movement control, balance, and functional mobility. Using dynamic surface for exercise provides proprioceptive and vestibular feedback about the position of their body segments in space with adaptive motor control response to stimuli. Standard physiotherapy based on motor-learning principle is task-specific training, which involves practice of functional movements in activities of daily living.

This study aims to describe the comparative effects of dynamic surface training and trunk targeted training in order to ensure which method is best in improving gross motor function , balance and trunk control in children with spastic cerebral palsy . this will be randomized control study which includes participants with age 5 to 10 years. Data will be taken from shahida islam teaching hospital Lodhran after taking consent, techniques will be applied and data will be recorded. Assessment will be made by using pedriatics balance scale , gross motor function measure (GMFM 66) and trunk control measurement scale (TCMS) for determining balance and gross motor function and trunk stability . The collective data will be analyzed in Statistical Package for Social Sciences (SPSS) 27.0

ELIGIBILITY:
Inclusion Criteria:

Children who can follow the therapist instructions

* Children who have not had any procedure and surgery within the past six months
* Both genders male and female
* Age 5 to 10 years
* Spastic cerebral palsy

Exclusion Criteria:

* Children with innate musculoskeletal diseases, developing Central nervous system diseases and history of orthopedic surgery

  * Children with genetic disorders and other severe diseases other than cerebral palsy
  * Children who had Botulinum Toxin A (BoNT-A) injection during the last 6 months or had seizures during the last one year were excluded from the study
  * Children with visual impairement
  * Children with hearing Impairemen

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-04-05 (Estimated); Study Completion 2023-04-05 (Estimated)

PRIMARY OUTCOMES:
pedriatic balance scale | 2 months
  Pediatric balance scale is an outcome measurement tool used to assess functional balance skills in children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points
gross motor function measure 88 GMFM-88 | 2 months
  The Gross Motor Function Measure (GMFM) is an observational clinical tool designed to evaluate change in gross motor function in children with cerebral palsy. There are two versions of the GMFM - the original 88-item measure (GMFM-88) and the more recent 66-item GMFM (GMFM-66). The scoring system of the GMFM is a four-point scale that consists of 66 items divided into five dimensions of gross motor function:(a) lying and rolling, (b) sitting, (c) crawling and kneeling, (d) standing, and (e) walking, running and jumping
Trunk control measurement scale | 2 months
  Trunk Control Measurement Scale is the clinical tool to measure trunk control in children with cerebral palsy. Control of muscles is necessary to maintain stability around the trunk.

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Altaf, Mphill, Principal Investigator — Riphah International University
Locations (1):
- Shahida Islam Teaching Hospital, Lodhran, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No